CLINICAL TRIAL: NCT02041806
Title: The Effectiveness of Peripheral Nerve Block Scoring Systems in Predicting the Success of a Block for Intra-Operative and Post-Operative Analgesia
Brief Title: Assessing Peripheral Nerve Block Scoring Systems for Intra-Operative and Post-Operative Analgesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Adelaide and Meath Hospital (Other)
Responsible Party: Principal Investigator, Dr Patrick Conroy, Consultant Anaesthesia, The Adelaide and Meath Hospital
Other Study IDs: SS/2013/81
Record Dates: First submitted 2014-01-16; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Complication of Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if Peripheral Nerve Block scoring systems are effective in predicting the achievement of intra-operative anaesthesia and post-operative analgesia.

DETAILED DESCRIPTION:
Upper and lower extremity surgery is particularly suited to regional anaesthesia. Peripheral nerve blocks (PNB) can produce surgical anaesthesia in less than 30 minutes. PNBs have been associated with early outcome improvements when surgery is conducted awake or with light sedation. These benefits include reduced nausea and vomiting, improved patient satisfaction and accelerated recovery room and hospital discharge. PNBs can also provide effective postoperative pain relief.

Currently there is no globally accepted standard by which to assess when surgical anaesthesia has been achieved following administration of PNBs. The decision as to when adequate surgical anaesthesia has been achieved and when surgery can then proceed is usually left to the discretion of the anaesthetist. The anaesthetist can assess nerve blockade though several motor and sensory function tests: cold, heat, touch and pinprick sensitivity. Several scoring systems have been described using these tests to estimate when surgical anaesthesia has been achieved but none have been independently validated outside of the original studies in which they have been described.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Grade I-IV

Exclusion Criteria:

* Contraindications to regional anesthesia
* Language barrier
* Existence of neurologic disease affecting the operative site
* Severe psychiatric disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing orthopaedic or vascular surgery who would receive a peripheral nerve block as part of their care.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Predictive value of block assessment score | 30 mins post block completion

CONTACTS AND LOCATIONS:
Overall Officials: Patrick H Conroy, Principal Investigator — The Adelaide and Meath Hospital
Locations (1):
- Tallaght Hospital, Dublin, Ireland